CLINICAL TRIAL: NCT02863575
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY COMPARING THE ANALGESIC EFFICACY AND SAFETY OF A SINGLE ORAL DOSE OF A NOVEL FIXED-DOSE COMBINATION OF IBUPROFEN 400 MG WITH CAFFEINE 100 MG TO IBUPROFEN 400 MG AND TO PLACEBO IN THE TREATMENT OF POST-SURGICAL DENTAL PAIN IN OTHERWISE HEALTHY SUBJECTS
Brief Title: A Dental Pain Study Comparing The Analgesic Efficacy Of Ibuprofen/Caffeine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B3741002; MIG (Other: Alias Study Number); MIG II (Other: Alias Study Number)
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Pain
Keywords: third molar extraction; ibuprofen; ibuprofen/caffeine; post-surgical dental pain
MeSH Terms: conditions — Pain | interventions — Ibuprofen; Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ibuprofen/Caffeine (Experimental): Ibuprofen 400 mg/ Caffeine 100 mg fixed-dose combination
  Interventions: Drug: Ibuprofen/Caffeine
- Ibuprofen (Active Comparator): Ibuprofen 400 mg
  Interventions: Drug: Ibuprofen
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen/Caffeine — Ibuprofen/Caffeine fixed-dose combination
  Arms: Ibuprofen/Caffeine
Drug: Ibuprofen — Ibuprofen capsule
  Arms: Ibuprofen
Drug: Placebo — Placebo treatment
  Arms: Placebo

SUMMARY:
An efficacy study assessing analgesic effect of ibuprofen/caffeine in post-surgical dental pain.

DETAILED DESCRIPTION:
The purpose of this study is to assess the analgesic efficacy of a fixed dose combination of ibuprofen/caffeine compared to ibuprofen alone and also to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 16 years to 40 years of age (inclusive).
* Subjects who have undergone outpatient surgical extraction of 3 or more third molars, of which at least 2 must be a partial or complete bony mandibular impaction within 30 days of Screening and have met baseline pain criteria as described in this protocol
* Examined by the attending dentist or physician and medically cleared to participate in the study.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, metabolic or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing) determined by the Investigator to place the subject at increased risk including the presence or history within 2 years of screening of the following medical conditions/disorders:

  * Bleeding disorder;
  * Gastrointestinal ulcer or gastrointestinal bleeding;
  * Paralytic ileus or other gastrointestinal obstructive disorders.
* Pregnant female subjects; breastfeeding female subjects; fertile male subjects and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception
* Hypersensitivity to ibuprofen, naproxen, aspirin, or any other NSAID, caffeine, or other component of the product.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 374 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3741002&StudyName=A+Phase+3%2C+Randomized%2C+Double-blind%2C+Placebo-controlled+Study+Comparing+The+Analgesic+Efficacy+And+Safety+Of+A+Single+Oral+Dose+Of+A+Novel+Fixed-dose+Combination+Of+Ibuprofen+400+Mg+With+Caffeine+100+Mg+To+Ibuprofen+400+Mg+And+To+Placebo+In+The+Treatment+Of+Post-surgical+Dental+Pain+In+Otherwise+Healthy+Subjects

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibuprofen 400 mg + Caffeine 100 mg: Participants were randomized to receive a single oral dose of ibuprofen 400 milligram (mg) with caffeine 100 mg as a fixed dose combination on Day 1. Participants were followed up to 17 days after the last dose of study drug.
- Ibuprofen 400 mg: Participants were randomized to receive a single oral dose of ibuprofen 400 mg on Day 1. Participants were followed up to 17 days after the last dose of study drug.
- Placebo: Participants were randomized to receive a single oral dose of Placebo (matched to ibuprofen 400 mg with caffeine 100 mg fixed dose combination) on Day 1. Participants were followed up to 17 days after the last dose of study drug.
Period: Overall Study
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg | Placebo
Started | 161 | 161 | 52
Completed | 160 | 159 | 51
Not Completed | 1 | 2 | 1
Not completed — Participants Unable To Swallow Capsule | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received the study medication.
Groups:
- Ibuprofen 400 mg + Caffeine 100 mg: Participants were randomized to receive a single oral dose of ibuprofen 400 mg with caffeine 100 mg as a fixed dose combination on Day 1. Participants were followed up to 17 days after the last dose of study drug.
- Total: Total of all reporting groups
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg | Placebo | Total
Number analyzed (Participants) | 161 | 161 | 52 | 374
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.3 (3.03) | 19.1 (2.88) | 18.9 (2.93) | 19.1 (2.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 84 | 27 | 196
  Male | 76 | 77 | 25 | 178
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 26 | 8 | 53
  Not Hispanic or Latino | 142 | 135 | 44 | 321
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 153 | 142 | 51 | 346
  Asian | 2 | 3 | 0 | 5
  Black or African American | 2 | 2 | 0 | 4
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 7 | 0 | 8
  Other | 2 | 6 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Time Weighted Sum of Pain Relief Rating (PRR) and Pain Intensity Difference (PID) Scores From 0 to 8 Hours Post-dose (SPRID 0-8): Ibuprofen + Caffeine Versus Ibuprofen
Description: SPRID 0-8: time-weighted sum of PRID scores from 0 to 8 hours. PRID: sum of PID and PRR at each post-dose time point. PRR score: at each post-dose time point participants answered to question "How much relief do you have from your starting pain?" on a 5-point scale: 0= none, 1= a little, 2= some, 3= a lot, 4= complete; higher scores = more relief from pain. Numerical pain severity rating (NPSR) scale: at baseline and each post-dose time point participants answered to question "How much pain do you have at this time?" on an 11-point scale: range from 0= no pain to 10= worst possible pain; higher scores = worse pain. PID score: NPSR score at baseline (0 hour) minus NPSR score at each post-dose time point; overall possible PID score range at a post-dose time point: -10 to 10, higher positive value = greater improvement. Overall possible SPRID 0-8 score range: -80 to 112, higher scores = more improvement in pain.
Time Frame: From 0 to 8 hours post-dose on Day 1
Population: Full analysis set (FAS) population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg
Number analyzed (Participants) | 161 | 161
units on a scale | 55.5 (1.8) | 52.8 (1.8)
Statistical Analysis 1: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; Test type: Superiority; p = 0.306, ANCOVA; Least square (LS) means difference = 2.68, 95% CI 2-sided [-2.46 to 7.82]

2. Secondary Outcome: Time Weighted Sum of Pain Relief Rating and Pain Intensity Difference Scores From 0 to 2 (SPRID 0-2), 0 to 4 (SPRID 0-4), 0 to 6 (SPRID 0-6) and 0 to 8 Hours Post-dose (SPRID 0-8)
Description: SPRID 0-2, SPRID 0-4, SPRID 0-6, SPRID 0-8: time-weighted sum of PRID scores from 0 to 2, 0 to 4, 0 to 6 and 0 to 8 hours respectively. PRID at each post-dose time point = PID + PRR. PRR score: at each post-dose time point participants answered to question "How much relief do you have from your starting pain?" on 5-point scale: 0=none, 1=a little, 2=some, 3=a lot, 4=complete; higher scores=more relief from pain. NPSR scale: at baseline and each post-dose time point participants answered to question "How much pain do you have at this time?" on 11-point scale: range from 0=no pain to 10=worst possible pain; higher scores=worse pain. PID score: NPSR score at baseline (0 hour) minus NPSR score at each post-dose time point; overall possible PID score range at a post-dose time point: -10 to 10, higher positive value=greater improvement. Score range for: SPRID 0-2= -20 to 28; SPRID 0-4= -40 to 56; SPRID 0-6= -60 to 84; SPRID 0-8= -80 to 112. Higher SPRID scores=more improvement in pain.
Time Frame: From 0 to 2, 0 to 4, 0 to 6 and 0 to 8 hours post-dose on Day 1
Population: FAS population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 161 | 161 | 52
units on a scale
  SPRID 0-2 | 13.3 (0.4) | 12.2 (0.4) | 2.2 (0.7)
  SPRID 0-4 | 30.0 (0.8) | 28.5 (0.8) | 6.0 (1.5)
  SPRID 0-6 | 44.5 (1.3) | 42.1 (1.3) | 10.2 (2.3)
  SPRID 0-8 | 55.5 (1.8) | 52.8 (1.8) | 14.6 (3.3)
Statistical Analysis 1: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; SPRID 0-2; Test type: Superiority; p = 0.056, ANCOVA; LS mean difference = 1.09, 95% CI 2-sided [-0.03 to 2.20]
Statistical Analysis 2: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; SPRID 0-2; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 11.13, 95% CI 2-sided [9.54 to 12.73]
Statistical Analysis 3: Comparison: Ibuprofen 400 mg vs Placebo; SPRID 0-2; Test type: Superiority; p < 0.001, ANCOVA; LS mean difference = 10.05, 95% CI 2-sided [8.45 to 11.64]
Statistical Analysis 4: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; SPRID 0-4; Test type: Superiority; p = 0.177, ANCOVA; LS mean difference = 1.58, 95% CI 2-sided [-0.72 to 3.87]
Statistical Analysis 5: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; SPRID 0-4; Test type: Superiority; p < 0.001, ANCOVA; LS mean difference = 24.04, 95% CI 2-sided [20.76 to 27.32]
Statistical Analysis 6: Comparison: Ibuprofen 400 mg vs Placebo; SPRID 0-4; Test type: Superiority; p < 0.001, ANCOVA; LS mean difference = 22.46, 95% CI 2-sided [19.18 to 25.75]
Statistical Analysis 7: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; SPRID 0-6; Test type: Superiority; p = 0.201, ANCOVA; LS mean difference = 2.39, 95% CI 2-sided [-1.28 to 6.06]
Statistical Analysis 8: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; SPRID 0-6; Test type: Superiority; p < 0.001, ANCOVA; LS mean difference = 34.30, 95% CI 2-sided [29.06 to 39.55]
Statistical Analysis 9: Comparison: Ibuprofen 400 mg vs Placebo; SPRID 0-6; Test type: Superiority; p < 0.001, ANCOVA; LS mean difference = 31.91, 95% CI 2-sided [26.67 to 37.16]
Statistical Analysis 10: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; SPRID 0-8; Test type: Superiority; p < 0.001, ANCOVA; LS mean difference = 40.85, 95% CI 2-sided [33.49 to 48.20]
Statistical Analysis 11: Comparison: Ibuprofen 400 mg vs Placebo; SPRID 0-8; Test type: Superiority; p < 0.001, ANCOVA; LS mean difference = 38.17, 95% CI 2-sided [30.81 to 45.52]

3. Secondary Outcome: Time Weighted Sum of Pain Intensity Difference Scores From 0 to 2 Hours (SPID 0-2), 0 to 4 (SPID 0-4), 0 to 6 (SPID 0-6) and 0 to 8 Hours Post-dose (SPID 0-8)
Description: SPID 0-2, SPID 0-4, SPID 0-6, SPID 0-8: time-weighted sum of PID scores from 0 to 2, 0 to 4, 0 to 6 and 0 to 8 hours post-dose respectively. NPSR scale: at baseline and each post-dose time point participants answered to question "How much pain do you have at this time?" on an 11-point scale: score range from 0 = no pain to 10 = worst possible pain; higher scores = worse pain. PID score: NPSR score at baseline (0 hour) minus NPSR score at each post-dose time point; overall possible PID score range at a post-dose time point: -10 to 10, higher positive value = greater improvement. Overall possible range: SPID 0-2 = -20 to 20; SPID 0-4 = -40 to 40; SPID 0-6 = -60 to 60; SPID 0-8 = -80 to 80. Higher SPID scores = more improvement in pain.
Time Frame: From 0 to 2, 0 to 4, 0 to 6 and 0 to 8 hours post-dose on Day 1
Population: FAS population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 161 | 161 | 52
units on a scale
  SPID 0-2 | 8.7 (0.3) | 8.0 (0.3) | 1.2 (0.5)
  SPID 0-4 | 19.9 (0.6) | 18.8 (0.6) | 3.5 (1.0)
  SPID 0-6 | 29.5 (0.9) | 27.7 (0.9) | 6.1 (1.6)
  SPID 0-8 | 36.6 (1.3) | 34.6 (1.3) | 8.8 (2.3)
Statistical Analysis 1: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; SPID 0-2; Test type: Superiority; p = 0.066, ANCOVA; LS means difference = 0.73, 95% CI 2-sided [-0.05 to 1.50]
Statistical Analysis 2: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; SPID 0-2; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 7.55, 95% CI 2-sided [6.44 to 8.66]
Statistical Analysis 3: Comparison: Ibuprofen 400 mg vs Placebo; SPID 0-2; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 6.82, 95% CI 2-sided [5.71 to 7.93]
Statistical Analysis 4: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; SPID 0-4; Test type: Superiority; p = 0.165, ANCOVA; LS means difference = 1.14, 95% CI 2-sided [-0.47 to 2.74]
Statistical Analysis 5: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; SPID 0-4; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 16.35, 95% CI 2-sided [14.05 to 18.64]
Statistical Analysis 6: Comparison: Ibuprofen 400 mg vs Placebo; SPID 0-4; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 15.21, 95% CI 2-sided [12.91 to 17.51]
Statistical Analysis 7: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; SPID 0-6; Test type: Superiority; p = 0.172, ANCOVA; LS means difference = 1.78, 95% CI 2-sided [-0.78 to 4.34]
Statistical Analysis 8: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; SPID 0-6; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 23.37, 95% CI 2-sided [19.71 to 27.03]
Statistical Analysis 9: Comparison: Ibuprofen 400 mg vs Placebo; SPID 0-6; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 21.59, 95% CI 2-sided [17.93 to 25.25]
Statistical Analysis 10: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; SPID 0-8; Test type: Superiority; p = 0.249, ANCOVA; LS means difference = 2.10, 95% CI 2-sided [-1.47 to 5.67]
Statistical Analysis 11: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; SPID 0-8; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 27.88, 95% CI 2-sided [22.78 to 32.99]
Statistical Analysis 12: Comparison: Ibuprofen 400 mg vs Placebo; SPID 0-8; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 25.79, 95% CI 2-sided [20.68 to 30.89]

4. Secondary Outcome: Time Weighted Sum of Pain Relief Rating Scores From 0 to 2 (TOTPAR 0-2), 0 to 4 (TOTPAR 0-4), 0 to 6 (TOTPAR 0-6) and 0 to 8 Hours Post-dose (TOTPAR 0-8)
Description: TOTPAR 0-2, TOTPAR 0-4, TOTPAR 0-6, TOTPAR 0-8: time-weighted sum of PRR scores from 0 to 2, 0 to 4, 0 to 6 and 0 to 8 hours post-dose respectively. PRR score: at each post-dose time point participants answered to the question "How much relief do you have from your starting pain?" on a 5-point scale: 0= none, 1= a little, 2= some, 3= a lot, 4= complete; higher scores = more relief from pain. Overall possible range: TOTPAR 0-2 = 0 to 8; TOTPAR 0-4 = 0 to 16; TOTPAR 0-6 = 0 to 24; TOTPAR 0-8 = 0 to 32. Higher TOTPAR scores = more improvement in pain.
Time Frame: From 0 to 2, 0 to 4, 0 to 6 and 0 to 8 hours post-dose on Day 1
Population: FAS population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 161 | 161 | 52
units on a scale
  TOTPAR 0-2 | 4.6 (0.1) | 4.2 (0.1) | 1.0 (0.2)
  TOTPAR 0-4 | 10.2 (0.3) | 9.7 (0.3) | 2.5 (0.5)
  TOTPAR 0-6 | 15.0 (0.4) | 14.4 (0.4) | 4.1 (0.7)
  TOTPAR 0-8 | 18.8 (0.6) | 18.2 (0.6) | 5.8 (1.0)
Statistical Analysis 1: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; TOTPAR 0-2; Test type: Superiority; p = 0.044, ANCOVA; LS means difference = 0.36, 95% CI 2-sided [0.01 to 0.71]
Statistical Analysis 2: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; TOTPAR 0-2; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 3.59, 95% CI 2-sided [3.09 to 4.09]
Statistical Analysis 3: Comparison: Ibuprofen 400 mg vs Placebo; TOTPAR 0-2; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 3.23, 95% CI 2-sided [2.73 to 3.73]
Statistical Analysis 4: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; TOTPAR 0-4; Test type: Superiority; p = 0.224, ANCOVA; LS means difference = 0.44, 95% CI 2-sided [-0.27 to 1.15]
Statistical Analysis 5: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; TOTPAR 0-4; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 7.69, 95% CI 2-sided [6.68 to 8.71]
Statistical Analysis 6: Comparison: Ibuprofen 400 mg vs Placebo; TOTPAR 0-4; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 7.25, 95% CI 2-sided [6.23 to 8.27]
Statistical Analysis 7: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; TOTPAR 0-6; Test type: Superiority; p = 0.293, ANCOVA; LS means difference = 0.61, 95% CI 2-sided [-0.53 to 1.75]
Statistical Analysis 8: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; TOTPAR 0-6; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 10.93, 95% CI 2-sided [9.30 to 12.56]
Statistical Analysis 9: Comparison: Ibuprofen 400 mg vs Placebo; TOTPAR 0-6; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 10.32, 95% CI 2-sided [8.69 to 11.95]
Statistical Analysis 10: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; TOTPAR 0-8; Test type: Superiority; p = 0.476, ANCOVA; LS means difference = 0.58, 95% CI 2-sided [-1.03 to 2.19]
Statistical Analysis 11: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; TOTPAR 0-8; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 12.96, 95% CI 2-sided [10.66 to 15.26]
Statistical Analysis 12: Comparison: Ibuprofen 400 mg vs Placebo; TOTPAR 0-8; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 12.38, 95% CI 2-sided [10.08 to 14.68]

5. Secondary Outcome: Sum of Pain Relief Rating and Pain Intensity Difference (PRID) Scores at 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, and 8 Hours Post-dose
Description: PRID: sum of PID and PRR at each post-dose time point. PRR score: at each post-dose time point participants answered to a question "How much relief do you have from your starting pain?" on a 5-point scale: 0= none, 1= a little, 2= some, 3= a lot, 4= complete; higher scores = more relief from pain. NPSR scale: at baseline and each post-dose time point participants answered to a question "How much pain do you have at this time?" on an 11-point scale: range from 0= no pain to 10= worst possible pain; higher scores = worse pain. PID score: NPSR score at baseline (0 hour) minus NPSR score at each post-dose time point; overall possible PID score range at a post-dose time point: -10 to 10, higher positive value = greater improvement. At a single post-dose time point overall possible range for PRID score: -10 to 14, higher scores = more improvement in pain.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, and 8 hours post-dose on Day 1
Population: FAS population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 161 | 161 | 52
units on a scale
  0.25 hour | 0.8 (0.1) | 0.8 (0.1) | 0.7 (0.2)
  0.5 hour | 3.3 (0.2) | 3.3 (0.2) | 1.0 (0.4)
  1 hour | 7.2 (0.2) | 6.5 (0.2) | 1.1 (0.4)
  1.5 hour | 8.5 (0.2) | 7.7 (0.2) | 1.1 (0.4)
  2 hour | 8.9 (0.2) | 8.3 (0.2) | 1.3 (0.4)
  3 hour | 8.7 (0.2) | 8.3 (0.2) | 1.8 (0.4)
  4 hour | 8.1 (0.3) | 8.0 (0.3) | 2.0 (0.5)
  5 hour | 7.6 (0.3) | 7.3 (0.3) | 2.1 (0.5)
  6 hour | 6.9 (0.3) | 6.4 (0.3) | 2.1 (0.5)
  7 hour | 5.7 (0.3) | 5.6 (0.3) | 2.2 (0.6)
  8 hour | 5.2 (0.3) | 5.0 (0.3) | 2.2 (0.6)
Statistical Analysis 1: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRID at 0.25 hour; Test type: Superiority; p = 0.975, ANCOVA; LS means difference = 0.01, 95% CI 2-sided [-0.35 to 0.36]
Statistical Analysis 2: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRID at 0.25 hour; Test type: Superiority; p = 0.654, ANCOVA; LS means difference = 0.12, 95% CI 2-sided [-0.40 to 0.63]
Statistical Analysis 3: Comparison: Ibuprofen 400 mg vs Placebo; PRID at 0.25 hour; Test type: Superiority; p = 0.670, ANCOVA; LS means difference = 0.11, 95% CI 2-sided [-0.40 to 0.62]
Statistical Analysis 4: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRID at 0.5 hour; Test type: Superiority; p = 0.917, ANCOVA; LS means difference = -0.04, 95% CI 2-sided [-0.70 to 0.63]
Statistical Analysis 5: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRID at 0.5 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 2.26, 95% CI 2-sided [1.31 to 3.20]
Statistical Analysis 6: Comparison: Ibuprofen 400 mg vs Placebo; PRID at 0.5 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 2.29, 95% CI 2-sided [1.35 to 3.24]
Statistical Analysis 7: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRID at 1 hour; Test type: Superiority; p = 0.039, ANCOVA; LS means difference = 0.73, 95% CI 2-sided [0.04 to 1.42]
Statistical Analysis 8: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRID at 1 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 6.11, 95% CI 2-sided [5.12 to 7.10]
Statistical Analysis 9: Comparison: Ibuprofen 400 mg vs Placebo; PRID at 1 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 5.38, 95% CI 2-sided [4.39 to 6.37]
Statistical Analysis 10: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRID at 1.5 hour; Test type: Superiority; p = 0.015, ANCOVA; LS means difference = 0.84, 95% CI 2-sided [0.16 to 1.52]
Statistical Analysis 11: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRID at 1.5 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 7.36, 95% CI 2-sided [6.39 to 8.33]
Statistical Analysis 12: Comparison: Ibuprofen 400 mg vs Placebo; PRID at 1.5 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 6.52, 95% CI 2-sided [5.55 to 7.49]
Statistical Analysis 13: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRID at 2 hour; Test type: Superiority; p = 0.071, ANCOVA; LS means difference = 0.62, 95% CI 2-sided [-0.05 to 1.30]
Statistical Analysis 14: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRID at 2 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 7.62, 95% CI 2-sided [6.65 to 8.58]
Statistical Analysis 15: Comparison: Ibuprofen 400 mg vs Placebo; PRID at 2 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 6.99, 95% CI 2-sided [6.03 to 7.96]
Statistical Analysis 16: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRID at 3 hour; Test type: Superiority; p = 0.243, ANCOVA; LS means difference = 0.41, 95% CI 2-sided [-0.28 to 1.09]
Statistical Analysis 17: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRID at 3 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 6.83, 95% CI 2-sided [5.85 to 7.80]
Statistical Analysis 18: Comparison: Ibuprofen 400 mg vs Placebo; PRID at 3 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 6.42, 95% CI 2-sided [5.44 to 7.40]
Statistical Analysis 19: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRID at 4 hour; Test type: Superiority; p = 0.823, ANCOVA; LS means difference = 0.08, 95% CI 2-sided [-0.65 to 0.82]
Statistical Analysis 20: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRID at 4 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 6.08, 95% CI 2-sided [5.02 to 7.14]
Statistical Analysis 21: Comparison: Ibuprofen 400 mg vs Placebo; PRID at 4 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 6.00, 95% CI 2-sided [4.94 to 7.05]
Statistical Analysis 22: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRID at 5 hour; Test type: Superiority; p = 0.438, ANCOVA; LS means difference = 0.31, 95% CI 2-sided [-0.48 to 1.11]
Statistical Analysis 23: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRID at 5 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 5.47, 95% CI 2-sided [4.33 to 6.60]
Statistical Analysis 24: Comparison: Ibuprofen 400 mg vs Placebo; PRID at 5 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 5.15, 95% CI 2-sided [4.01 to 6.29]
Statistical Analysis 25: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRID at 6 hour; Test type: Superiority; p = 0.250, ANCOVA; LS means difference = 0.50, 95% CI 2-sided [-0.35 to 1.35]
Statistical Analysis 26: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRID at 6 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 4.80, 95% CI 2-sided [3.58 to 6.02]
Statistical Analysis 27: Comparison: Ibuprofen 400 mg vs Placebo; PRID at 6 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 4.30, 95% CI 2-sided [3.08 to 5.52]
Statistical Analysis 28: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRID at 7 hour; Test type: Superiority; p = 0.818, ANCOVA; LS means difference = 0.11, 95% CI 2-sided [-0.80 to 1.01]
Statistical Analysis 29: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRID at 7 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 3.53, 95% CI 2-sided [2.23 to 4.82]
Statistical Analysis 30: Comparison: Ibuprofen 400 mg vs Placebo; PRID at 7 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 3.42, 95% CI 2-sided [2.12 to 4.71]
Statistical Analysis 31: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRID at 8 hour; Test type: Superiority; p = 0.698, ANCOVA; LS means difference = 0.18, 95% CI 2-sided [-0.74 to 1.11]
Statistical Analysis 32: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRID at 8 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 3.02, 95% CI 2-sided [1.69 to 4.34]
Statistical Analysis 33: Comparison: Ibuprofen 400 mg vs Placebo; PRID at 8 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 2.83, 95% CI 2-sided [1.51 to 4.16]

6. Secondary Outcome: Pain Relief Rating Scores at 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, and 8 Hours Post-dose
Description: PRR score: at each post-dose time point participants answered to a question "How much relief do you have from your starting pain?" on a 5-point scale: 0= none, 1= a little, 2= some, 3= a lot, 4= complete; higher scores = more relief from pain.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4 5, 6, 7, and 8 hours post-dose on Day 1
Population: FAS population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 161 | 161 | 52
units on a scale
  0.25 hour | 0.4 (0.0) | 0.4 (0.0) | 0.3 (0.1)
  0.5 hour | 1.3 (0.1) | 1.2 (0.1) | 0.5 (0.1)
  1 hour | 2.5 (0.1) | 2.3 (0.1) | 0.5 (0.1)
  1.5 hour | 2.8 (0.1) | 2.6 (0.1) | 0.5 (0.1)
  2 hour | 3.0 (0.1) | 2.8 (0.1) | 0.6 (0.1)
  3 hour | 2.9 (0.1) | 2.8 (0.1) | 0.7 (0.1)
  4 hour | 2.7 (0.1) | 2.7 (0.1) | 0.8 (0.1)
  5 hour | 2.6 (0.1) | 2.5 (0.1) | 0.8 (0.2)
  6 hour | 2.3 (0.1) | 2.2 (0.1) | 0.8 (0.2)
  7 hour | 2.0 (0.1) | 2.0 (0.1) | 0.9 (0.2)
  8 hour | 1.8 (0.1) | 1.8 (0.1) | 0.9 (0.2)
Statistical Analysis 1: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRR score at 0.25 hour; Test type: Superiority; p = 0.575, ANCOVA; LS means difference = 0.04, 94% CI 2-sided [-0.09 to 0.16]
Statistical Analysis 2: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRR score at 0.25 hour; Test type: Superiority; p = 0.426, ANCOVA; LS means difference = 0.07, 95% CI 2-sided [-0.11 to 0.25]
Statistical Analysis 3: Comparison: Ibuprofen 400 mg vs Placebo; PRR score at 0.25 hour; Test type: Superiority; p = 0.686, ANCOVA; LS means difference = 0.04, 95% CI 2-sided [-0.14 to 0.22]
Statistical Analysis 4: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRR score at 0.5 hour; Test type: Superiority; p = 0.543, ANCOVA; LS means difference = 0.07, 95% CI 2-sided [-0.15 to 0.29]
Statistical Analysis 5: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRR score at 0.5 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 0.81, 95% CI 2-sided [0.49 to 1.12]
Statistical Analysis 6: Comparison: Ibuprofen 400 mg vs Placebo; PRR score at 0.5 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 0.74, 95% CI 2-sided [0.42 to 1.05]
Statistical Analysis 7: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRR score at 1 hour; Test type: Superiority; p = 0.038, ANCOVA; LS means difference = 0.24, 95% CI 2-sided [0.01 to 0.46]
Statistical Analysis 8: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRR score at 1 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 2.01, 95% CI 2-sided [1.69 to 2.33]
Statistical Analysis 9: Comparison: Ibuprofen 400 mg vs Placebo; PRR score at 1 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 1.78, 95% CI 2-sided [1.46 to 2.09]
Statistical Analysis 10: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRR score at 1.5 hour; Test type: Superiority; p = 0.024, ANCOVA; LS means difference = 0.25, 95% CI 2-sided [0.03 to 0.47]
Statistical Analysis 11: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRR score at 1.5 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 2.33, 95% CI 2-sided [2.02 to 2.64]
Statistical Analysis 12: Comparison: Ibuprofen 400 mg vs Placebo; PRR score at 1.5 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 2.08, 95% CI 2-sided [1.77 to 2.39]
Statistical Analysis 13: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRR score at 2 hour; Test type: Superiority; p = 0.103, ANCOVA; LS means difference = 0.18, 95% CI 2-sided [-0.04 to 0.40]
Statistical Analysis 14: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRR score at 2 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 2.40, 95% CI 2-sided [2.09 to 2.71]
Statistical Analysis 15: Comparison: Ibuprofen 400 mg vs Placebo; PRR score at 2 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 2.22, 95% CI 2-sided [1.91 to 2.53]
Statistical Analysis 16: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRR score at 3 hour; Test type: Superiority; p = 0.448, ANCOVA; LS means difference = 0.08, 95% CI 2-sided [-0.13 to 0.29]
Statistical Analysis 17: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRR score at 3 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 2.16, 95% CI 2-sided [1.86 to 2.47]
Statistical Analysis 18: Comparison: Ibuprofen 400 mg vs Placebo; PRR score at 3 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 2.08, 95% CI 2-sided [1.78 to 2.38]
Statistical Analysis 19: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRR score at 4 hour; Test type: Superiority; p = 0.997, ANCOVA; LS means difference = 0.00, 95% CI 2-sided [-0.23 to 0.23]
Statistical Analysis 20: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRR score at 4 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 1.94, 95% CI 2-sided [1.61 to 2.28]
Statistical Analysis 21: Comparison: Ibuprofen 400 mg vs Placebo; PRR score at 4 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 1.94, 95% CI 2-sided [1.61 to 2.28]
Statistical Analysis 22: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRR score at 5 hour; Test type: Superiority; p = 0.656, ANCOVA; LS means difference = 0.06, 95% CI 2-sided [-0.19 to 0.31]
Statistical Analysis 23: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRR score at 5 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 1.73, 95% CI 2-sided [1.36 to 2.09]
Statistical Analysis 24: Comparison: Ibuprofen 400 mg vs Placebo; PRR score at 5 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 1.67, 95% CI 2-sided [1.31 to 2.03]
Statistical Analysis 25: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRR score at 6 hour; Test type: Superiority; p = 0.425, ANCOVA; LS means difference = 0.11, 94% CI 2-sided [-0.16 to 0.38]
Statistical Analysis 26: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRR score at 6 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 1.51, 95% CI 2-sided [1.12 to 1.90]
Statistical Analysis 27: Comparison: Ibuprofen 400 mg vs Placebo; PRR score at 6 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 1.40, 95% CI 2-sided [1.01 to 1.79]
Statistical Analysis 28: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRR score at 7 hour; Test type: Superiority; p = 0.841, ANCOVA; LS means difference = -0.03, 95% CI 2-sided [-0.32 to 0.26]
Statistical Analysis 29: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRR score at 7 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 1.10, 95% CI 2-sided [0.69 to 1.52]
Statistical Analysis 30: Comparison: Ibuprofen 400 mg vs Placebo; PRR score at 7 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 1.13, 95% CI 2-sided [0.72 to 1.55]
Statistical Analysis 31: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PRR score at 8 hour; Test type: Superiority; p = 0.980, ANCOVA; LS means difference = 0.00, 95% CI [-0.30 to 0.30]
Statistical Analysis 32: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PRR score at 8 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 0.93, 95% CI 2-sided [0.50 to 1.36]
Statistical Analysis 33: Comparison: Ibuprofen 400 mg vs Placebo; PRR score at 8 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 0.93, 95% CI 2-sided [0.50 to 1.35]

7. Secondary Outcome: Pain Intensity Difference Scores at 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, and 8 Hours Post-dose
Description: NPSR scale: at baseline and each post-dose time point participants answered to a question "How much pain do you have at this time?" on an 11-point scale: range from 0= no pain to 10= worst possible pain; higher scores = worse pain. PID score: NPSR score at baseline (0 hour) minus NPSR score at each post-dose time point; overall possible PID score range at a single post-dose time point: -10 to 10, higher positive value = greater improvement in pain.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4 5, 6, 7, and 8 hours post-dose on Day 1
Population: FAS population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 161 | 161 | 52
units on a scale
  0.25 hour | 0.4 (0.1) | 0.5 (0.1) | 0.4 (0.2)
  0.5 hour | 2.0 (0.2) | 2.1 (0.2) | 0.6 (0.3)
  1 hour | 4.7 (0.2) | 4.2 (0.2) | 0.6 (0.3)
  1.5 hour | 5.6 (0.2) | 5.1 (0.2) | 0.6 (0.3)
  2 hour | 5.9 (0.2) | 5.5 (0.2) | 0.7 (0.3)
  3 hour | 5.8 (0.2) | 5.5 (0.2) | 1.1 (0.3)
  4 hour | 5.4 (0.2) | 5.3 (0.2) | 1.2 (0.3)
  5 hour | 5.0 (0.2) | 4.8 (0.2) | 1.3 (0.3)
  6 hour | 4.5 (0.2) | 4.1 (0.2) | 1.2 (0.4)
  7 hour | 3.8 (0.2) | 3.6 (0.2) | 1.3 (0.4)
  8 hour | 3.4 (0.2) | 3.3 (0.2) | 1.3 (0.4)
Statistical Analysis 1: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PID score at 0.25 hour; Test type: Superiority; p = 0.808, ANCOVA; LS means difference = -0.03, 95% CI 2-sided [-0.27 to 0.21]
Statistical Analysis 2: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PID score at 0.25 hour; Test type: Superiority; p = 0.804, ANCOVA; LS means difference = 0.04, 95% CI 2-sided [-0.30 to 0.39]
Statistical Analysis 3: Comparison: Ibuprofen 400 mg vs Placebo; PID score at 0.25 hr; Test type: Superiority; p = 0.676, ANCOVA; LS means difference = 0.07, 95% CI 2-sided [-0.27 to 0.42]
Statistical Analysis 4: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PID score at 0.5 hour; Test type: Superiority; p = 0.654, ANCOVA; LS means difference = -0.10, 95% CI 2-sided [-0.55 to 0.35]
Statistical Analysis 5: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PID score at 0.5 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 1.45, 95% CI 2-sided [0.81 to 2.10]
Statistical Analysis 6: Comparison: Ibuprofen 400 mg vs Placebo; PID score at 0.5 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 1.55, 95% CI 2-sided [0.91 to 2.20]
Statistical Analysis 7: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PID score at 1 hour; Test type: Superiority; p = 0.045, ANCOVA; LS means difference = 0.49, 95% CI 2-sided [0.01 to 0.97]
Statistical Analysis 8: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PID score at 1 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 4.10, 95% CI [3.41 to 4.78]
Statistical Analysis 9: Comparison: Ibuprofen 400 mg vs Placebo; PID score at 1 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 3.60, 95% CI 2-sided [2.92 to 4.29]
Statistical Analysis 10: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PID score at 1.5 hour; Test type: Superiority; p = 0.015, ANCOVA; LS means difference = 0.59, 95% CI 2-sided [0.11 to 1.06]
Statistical Analysis 11: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PID score at 1.5 hour; Test type: Superiority; p < 0.001, ANOVA; LS means difference = 5.03, 95% CI 2-sided [4.35 to 5.71]
Statistical Analysis 12: Comparison: Ibuprofen 400 mg vs Placebo; PID score at 1.5 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 4.44, 95% CI 2-sided [3.76 to 5.12]
Statistical Analysis 13: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PID score at 2 hour; Test type: Superiority; p = 0.066, ANCOVA; LS means difference = 0.44, 95% CI 2-sided [-0.03 to 0.91]
Statistical Analysis 14: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PID score at 2 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 5.22, 95% CI 2-sided [4.54 to 5.89]
Statistical Analysis 15: Comparison: Ibuprofen 400 mg vs Placebo; PID score at 2 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 4.78, 95% CI 2-sided [4.10 to 5.45]
Statistical Analysis 16: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PID score at 3 hour; Test type: Superiority; p = 0.186, ANCOVA; LS means difference = 0.32, 95% CI 2-sided [-0.16 to 0.81]
Statistical Analysis 17: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PID score at 3 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 4.66, 95% CI 2-sided [3.98 to 5.35]
Statistical Analysis 18: Comparison: Ibuprofen 400 mg vs Placebo; PID score at 3 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 4.34, 95% CI 2-sided [3.65 to 5.03]
Statistical Analysis 19: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PID score at 4 hour; Test type: Superiority; p = 0.750, ANCOVA; LS means difference = 0.08, 95% CI 2-sided [-0.43 to 0.60]
Statistical Analysis 20: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PID score at 4 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 4.14, 95% CI 2-sided [3.40 to 4.87]
Statistical Analysis 21: Comparison: Ibuprofen 400 mg vs Placebo; PID score at 4 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 4.05, 95% CI 2-sided [3.32 to 4.79]
Statistical Analysis 22: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PID score at 5 hour; Test type: Superiority; p = 0.361, ANCOVA; LS means difference = 0.26, 95% CI 2-sided [-0.30 to 0.81]
Statistical Analysis 23: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PID score at 5 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 3.74, 95% CI 2-sided [2.95 to 4.53]
Statistical Analysis 24: Comparison: Ibuprofen 400 mg vs Placebo; PID score at 5 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 3.48, 95% CI 2-sided [2.69 to 4.27]
Statistical Analysis 25: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PID score at 6 hour; Test type: Superiority; p = 0.195, ANCOVA; LS means difference = 0.39, 95% CI 2-sided [-0.20 to 0.98]
Statistical Analysis 26: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PID score at 6 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 3.29, 95% CI 2-sided [2.44 to 4.13]
Statistical Analysis 27: Comparison: Ibuprofen 400 mg vs Placebo; PID score at 6 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 2.90, 95% CI 2-sided [2.06 to 3.74]
Statistical Analysis 28: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PID score at 7 hour; Test type: Superiority; p = 0.669, ANCOVA; LS means difference = 0.14, 95% CI 2-sided [-0.49 to 0.76]
Statistical Analysis 29: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PID score at 7 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 2.42, 95% CI 2-sided [1.53 to 3.31]
Statistical Analysis 30: Comparison: Ibuprofen 400 mg vs Placebo; PID score at 7 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 2.29, 95% CI 2-sided [1.40 to 3.18]
Statistical Analysis 31: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; PID score at 8 hour; Test type: Superiority; p = 0.581, ANCOVA; LS means difference = 0.18, 95% CI 2-sided [-0.46 to 0.82]
Statistical Analysis 32: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; PID score at 8 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 2.09, 95% CI 2-sided [1.18 to 3.00]
Statistical Analysis 33: Comparison: Ibuprofen 400 mg vs Placebo; PID score at 8 hour; Test type: Superiority; p < 0.001, ANCOVA; LS means difference = 1.91, 95% CI 2-sided [1.00 to 2.82]

8. Secondary Outcome: Time to Onset of Achieving Meaningful Relief
Description: When the participants were administered study medication at time 0 hours they were given the 2 stopwatches: 1 stopwatch was labelled as "first perceptible relief" and another as "meaningful relief." Participants were instructed to stop the stopwatch labelled as "meaningful relief" at the moment when they first experienced meaningful relief, that is, when the relief from the pain was meaningful to them. The stopwatch remained active for 8 hours (until stopped by the participants, or until rescue medication was administered).
Time Frame: Up to 8 hours post-dose on Day 1
Population: FAS population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 161 | 161 | 52
minutes | 46.60 [42.82 to 49.15] | 52.25 [49.15 to 59.18] | NA [NA to NA] — Due to smaller number of participants with an event, median and 95% CI could not be calculated.
Statistical Analysis 1: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; Test type: Superiority; p = 0.028, Gehan-Wilcoxon test; P-value was calculated using the Gehan-Wilcoxon test, stratified by gender and baseline categorical pain severity terms
Statistical Analysis 2: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; Test type: Superiority; p < 0.001, Gehan-Wilcoxon test; P-value was calculated using the Gehan-Wilcoxon test, stratified by gender and baseline categorical pain severity terms
Statistical Analysis 3: Comparison: Ibuprofen 400 mg vs Placebo; Test type: Superiority; p < 0.001, Gehan-Wilcoxon test; P-value was calculated using the Gehan-Wilcoxon test, stratified by gender and baseline categorical pain severity terms

9. Secondary Outcome: Time to Onset of First Perceptible Relief
Description: When the participants were administered study medication at time 0 hours they were given the 2 stopwatches: 1 stopwatch was labelled as "first perceptible relief" and another as "meaningful relief." Participants were instructed to stop the stopwatch labelled as "first perceptible relief" at the moment when they first began to feel any pain relieving effect. It was when they first felt a little/noticeable pain relief. It did not mean that they felt completely better (though they might), but when they first felt any difference in pain that they had at present. The stopwatch remained active for 8 hours (until stopped by the participants, or until rescue medication was administered).
Time Frame: Up to 8 hours post-dose on Day 1
Population: FAS population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 161 | 161 | 52
minutes | 25.80 [21.93 to 29.42] | 24.52 [22.78 to 26.90] | NA [NA to NA] — Due to smaller number of participants with an event, median and 95% CI could not be calculated.
Statistical Analysis 1: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; Test type: Superiority; p = 0.861, Gehan-Wilcoxon test; P-value was calculated using the Gehan-Wilcoxon test, stratified by gender and baseline categorical pain severity terms
Statistical Analysis 2: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; Test type: Superiority; p < 0.001, Gehan-Wilcoxon test; P-value was calculated using the Gehan-Wilcoxon test, stratified by gender and baseline categorical pain severity terms
Statistical Analysis 3: Comparison: Ibuprofen 400 mg vs Placebo; Test type: Superiority; p < 0.001, Gehan-Wilcoxon test; P-value was calculated using the Gehan-Wilcoxon test, stratified by gender and baseline categorical pain severity terms

10. Secondary Outcome: Time to Treatment Failure
Description: Treatment failure was defined as time to first dose of rescue medication or study discontinuation of the participants due to lack of efficacy.
Time Frame: Up to 8 hours post dose on Day 1
Population: FAS population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 161 | 161 | 52
minutes | NA [NA to NA] — Due to smaller number of participants with an event, median and 95% CI could not be calculated. | NA [NA to NA] — Due to smaller number of participants with an event, median and 95% CI could not be calculated. | 310.00 [132.00 to 480.00]
Statistical Analysis 1: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Ibuprofen 400 mg; Test type: Superiority; p = 0.838, Gehan-Wilcoxon test; P-value was calculated using the Gehan-Wilcoxon test, stratified by gender and baseline categorical pain severity terms
Statistical Analysis 2: Comparison: Ibuprofen 400 mg + Caffeine 100 mg vs Placebo; Test type: Superiority; p < 0.001, Gehan-Wilcoxon test; P-value was calculated using the Gehan-Wilcoxon test, stratified by gender and baseline categorical pain severity terms
Statistical Analysis 3: Comparison: Ibuprofen 400 mg vs Placebo; Test type: Superiority; p < 0.001, Gehan-Wilcoxon test; P-value was calculated using the Gehan-Wilcoxon test, stratified by gender and baseline categorical pain severity terms

11. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) by Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pre-treatment state. AEs are classified according to severity in 3 categories as mild (did not interfere with participant's usual function), moderate (interfered to some extent with participant's usual function) and severe (interfered significantly with participant's usual function).
Time Frame: Screening up to Day 17 after the last dose of study drug (approximately maximum of 48 days)
Population: Safety analysis population included all participants who received the study medication. Here, "Overall Number of Participants Analyzed" were those participants who had at least 1 treatment emergent AEs.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 15 | 15 | 8
Participants
  Mild | 3 | 8 | 0
  Moderate | 12 | 7 | 8
  Severe | 0 | 0 | 0

12. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Treatment Related Adverse Events (AEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pre-treatment state. Relatedness of an AE to study drug was assessed by investigator.
Time Frame: Screening up to Day 17 after the last dose of study drug (approximately maximum of 48 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 15 | 15 | 8
Participants | 1 | 2 | 2

13. Other Pre Specified Outcome: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Vital signs included: heart rate, blood pressure, respiratory rate, and temperature. Normal range for the vital signs were: systolic blood pressure 90 to 140 millimeter of mercury (mmHg), diastolic blood pressure 60 to 90 mmHg, heart rate 50 to 110 beats per minute, respiratory rate 12 to 22 breaths per minute, and oral temperature 97.0 to 99.6 Fahrenheit (F). Value for vital signs outside the normal range was consider as abnormal. Clinical significance of vital signs abnormalities was determined at the investigator's discretion.
Time Frame: Screening up to Day 17 after the last dose of study drug (approximately maximum of 48 days)
Population: Safety analysis population included all participants who received the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 161 | 161 | 52
Participants | 0 | 0 | 0

14. Other Pre Specified Outcome: Number of Participants Who Used Concomitant Medications, and Rescue Medications
Description: Rescue medication: participants who did not experience adequate relief after the 1 hour (post study drug dose) evaluation were given tramadol hydrochloride 50 to 100 mg orally or codeine sulfate 15 to 60 mg orally, based on the discretion of the Investigator, as rescue medication. If needed, 2 additional doses of rescue medications based on the discretion of the Investigator at the study center was given. Total maximum dose of tramadol was 300 mg and of codeine sulfate was 180 mg. Concomitant medication: medication received by participant other than study medication and rescue medication.
Time Frame: Day 1
Population: Safety analysis population included all participants who received the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 161 | 161 | 52
Participants
  Concomitant Medications | 25 | 39 | 11
  Rescue Medications | 29 | 25 | 28

15. Other Pre Specified Outcome: Number of Participants Who Used Medications Prior to This Study
Description: In this outcome measure number of participants who were using any type of medications, prior to start of the study were reported.
Time Frame: At Screening
Population: Safety analysis population included all participants who received the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg | Placebo
Number analyzed (Participants) | 161 | 161 | 52
Participants | 161 | 161 | 52

ADVERSE EVENTS:
Time Frame: Screening up to Day 17 after the last dose of study drug (approximately maximum 48 days)
Description: Safety population.
Arm/Group | Ibuprofen 400 mg + Caffeine 100 mg | Ibuprofen 400 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/161 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/161 | 0/161 | 0/52
Other Adverse Events (participants affected / at risk) | 15/161 | 15/161 | 8/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibuprofen 400 mg + Caffeine 100 mg (N=161) | Ibuprofen 400 mg (N=161) | Placebo (N=52)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 7
Pain (General disorders) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 2 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 6
Alveolar osteitis (Infections and infestations) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results

DOCUMENTS (2):
  • Study Protocol (2016-07-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT02863575/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/75/NCT02863575/SAP_001.pdf